CLINICAL TRIAL: NCT03197870
Title: Phase 2 Double-Masked, Placebo-Controlled Study to Assess the Safety and Efficacy of Subcutaneously Administered AKB-9778 (Razuprotafib)15mg Once Daily or 15mg Twice Daily for 12 Months in Patients With Moderate to Severe Non-Proliferative Diabetic Retinopathy
Brief Title: The TIME-2b Study: A Study of AKB-9778 (Razuprotafib), a Novel Tie 2 Activator, in Patients With Non-Proliferative Diabetic Retinopathy (NPDR)
Acronym: TIME-2b
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EyePoint Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AKB-9778-CI-5001
Record Dates: First submitted 2017-06-22; First posted 2017-06-23 (Actual); Results first posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Nonproliferative Diabetic Retinopathy
MeSH Terms: interventions — AKB-9778

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AKB-9778 15mg Daily (Experimental): AKB-9778 15 mg (QD); To maintain masking, subjects will receive BID dosing with masked study medication administered as one dose of active and one dose of matching placebo
  Interventions: Drug: AKB-9778; Drug: Placebo
- AKB-9778 15mg Twice Daily (Experimental): AKB-9778 15 mg (BID)
  Interventions: Drug: AKB-9778
- Placebo Twice Daily (Placebo Comparator): Placebo Group: SC Phosphate-Buffered-Saline (PBS) (BID)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AKB-9778 — Subcutaneous AKB-9778 15mg
  Arms: AKB-9778 15mg Daily; AKB-9778 15mg Twice Daily
Drug: Placebo — Subcutaneous Placebo
  Arms: AKB-9778 15mg Daily; Placebo Twice Daily

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of subcutaneously administered AKB-9778 15mg once daily or 15mg twice daily for 12 months in patients with moderate to severe non-proliferative diabetic retinopathy (NPDR).

ELIGIBILITY:
Key Inclusion Criteria:

* Adults 18 through 80 years of age (inclusive)
* Subjects with moderate to very severe NPDR (ETDRS Level 43 - 53 inclusive)
* No evidence of central involved diabetic macular edema
* ETDRS best-corrected visual acuity letter score ≥ 70 (Snellen 20/40 or better)

Key Exclusion Criteria:

* Ocular disease other than DR that may cause substantial reduction in visual acuity, including iris neovascularization, retinal detachment, visually significant epiretinal membrane, vitreous hemorrhage or fibrosis, ocular inflammation (uveitis), other retinal inflammatory or infectious diseases
* Evidence of neovascularization on clinical examination or imaging
* Hemoglobin A1C (HbA1C) ≥ 12.0% at Screening
* Severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-02-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (53):
- United States (53):
  - Arizona Retina and Vitreous Consultants, Phoenix, Arizona
  - Retinal Research Institute, Phoenix, Arizona
  - Retina Institute of California, Arcadia, California
  - California Retina Consultants, Bakersfield, California
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - Retina Consultants of Orange County, Fullerton, California
  - Ophthalmic Clinical Trials San Diego, Oceanside, California
  - Stanford, Palo Alto, California
  - California Retina Consultants, Santa Barbara, California
  - California Retina Consultants, Santa Maria, California
  - Retina Consultants of Southern Colorado, Colorado Springs, Colorado
  - Colorado Retina Associates, Golden, Colorado
  - Rand Eye Institute, Deerfield Beach, Florida
  - Center for Retina and Macular Disease, Lakeland, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina, Marietta, Georgia
  - University Retina, Oak Forest, Illinois
  - Illinois Retina Associates, Oak Park, Illinois
  - Midwest Eye Institute, Indianapolis, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Central Plains Eye MDs, Wichita, Kansas
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Cumberland Valley Retina Consultants PC, Hagerstown, Maryland
  - Opthalmic Consultants of Boston, Boston, Massachusetts
  - Specialty Eye Institute, Jackson, Michigan
  - Sierra Eye Associates, Reno, Nevada
  - Retina Center of New Jersey, Bloomfield, New Jersey
  - New Jersey Retina, Edison, New Jersey
  - Retinal and Ophthalmic Consultants P.C., Northfield, New Jersey
  - Eye Associates of New Mexico, Albuquerque, New Mexico
  - Island Retina, Shirley, New York
  - Retina Vitreous Surgeons of Central New York, Syracuse, New York
  - Retina Associates of Cleveland, Beachwood, Ohio
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Retina Associates of Cleveland, Middleburg Heights, Ohio
  - Retina Associates of Cleveland, Youngstown, Ohio
  - Retina Vitreous Center, Edmond, Oklahoma
  - Mid-Atlantic Retina, Bethlehem, Pennsylvania
  - Tennessee Retina, Nashville, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Texas Retina Associates, Arlington, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Research Center, Austin, Texas
  - Texas Retina Associates, Fort Worth, Texas
  - Valley Retina Institute, Harlingen, Texas
  - Retina and Vitreous of Texas, Houston, Texas
  - Retina Consultants of Houston, Houston, Texas
  - Valley Retina Institute, McAllen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - Spokane Eye Clinical Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Razuprotafib 15mg Twice Daily: Razuprotafib: Subcutaneous Razuprotafib 15mg
- Razuprotafib 15mg Daily: Razuprotafib: Subcutaneous Razuprotafib 15mg
  Placebo: Subcutaneous Placebo
Period: Overall Study
Arm/Group | Razuprotafib 15mg Twice Daily | Razuprotafib 15mg Daily | Placebo Twice Daily
Started | 55 | 55 | 57
Completed | 41 | 45 | 51
Not Completed | 14 | 10 | 6
Not completed — Adverse Event | 9 | 4 | 6
Not completed — Withdrawal by Subject | 2 | 3 | 0
Not completed — Lost to Follow-up | 2 | 2 | 0
Not completed — data not available | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Razuprotafib 15mg Twice Daily | Razuprotafib 15mg Daily | Placebo Twice Daily | Total
Number analyzed (Participants) | 55 | 55 | 57 | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (11.17) | 58.5 (10.69) | 55.9 (9.88) | 57.0 (10.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 25 | 71
  Male | 32 | 32 | 32 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 20 | 25 | 70
  Not Hispanic or Latino | 30 | 35 | 32 | 97
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Native Alaskan | 1 | 0 | 2 | 3
  Asian | 2 | 3 | 1 | 6
  Black/African American | 4 | 7 | 3 | 14
  Native Hawaiian/Pacific Islander | 0 | 0 | 1 | 1
  White | 47 | 45 | 49 | 141
  Other | 1 | 0 | 1 | 2
Body Mass Index, kg/m² [Mean (Standard Deviation); unit: kg/m²] | 31.91 (4.776) | 29.63 (5.138) | 30.58 (4.752) | 30.71 (4.949)
Hemoglobin A1c, % [Mean (Standard Deviation); unit: % of Glycated hemoglobin] | 8.58 (1.380) | 8.31 (1.885) | 8.18 (1.457) | 8.35 (1.587)
Type of Diabetes, n (%) [Count of Participants; unit: Participants]
  Type 1 | 6 | 6 | 4 | 16
  Type 2 | 49 | 49 | 53 | 151
Duration of Diabetes, years [Mean (Standard Deviation); unit: years] | 17.83 (12.232) | 17.78 (11.001) | 14.54 (8.625) | 16.69 (10.749)
Taking Insulin, n (%) [Count of Participants; unit: Participants]
  Yes | 43 | 37 | 33 | 113
  No | 12 | 18 | 24 | 54
Taking Angiotensin-Converting Enzyme Inhibitor (ACEi)/Angiotensin Receptor Blocker (ARB) [Count of Participants; unit: Participants]
  Yes | 29 | 39 | 33 | 101
  No | 26 | 16 | 24 | 66
Study eye, n (%) [Count of Participants; unit: Participants]
  Right Eye | 27 | 32 | 26 | 85
  Left Eye | 28 | 23 | 31 | 82
Duration of non-proliferative diabetic retinopathy in Study Eye, years [Mean (Standard Deviation); unit: years] — Population: The "n" for this Baseline Characteristic does not match the overall population. The overall number of participants analyzed represents the total number of participants in each treatment group for the safety population. The summary included only those participants with available data.
  years
    number analyzed (Participants) | 51 | 51 | 54 | 156
    (all) | 2.69 (4.360) | 2.04 (2.679) | 2.55 (4.267) | 2.43 (3.841)
Duration of NPDR in qualified fellow eye, years [Mean (Standard Deviation); unit: years] — If both eyes met all ocular eligibility criteria, then the eye with the worse ETDRS DRSS was designated the study eye, and the other eye designated as a qualified fellow eye; in this case, the Central Image Reading Center confirmed selection of the study eye. Not all subjects had a qualified fellow eye with NPDR (Non-Proliferative Diabetic Retinopathy). Population: Qualified fellow eyes only
  years
    number analyzed (Participants) | 13 | 17 | 20 | 50
    (all) | 1.78 (2.540) | 2.00 (3.282) | 2.14 (2.512) | 2.00 (2.750)
Prior Treatment for Proliferative Diabetic Retinopathy or Diabetic Macular Edema in Study Eye [Count of Participants; unit: Participants]
  Yes | 14 | 7 | 7 | 28
  No | 41 | 48 | 50 | 139
Prior Treatment for PDR or DME in Qualified Fellow Eye [Count of Participants; unit: Participants] — Population: If both eyes met all ocular eligibility criteria, then the eye with the worse ETDRS DRSS was designated the study eye, and the other eye designated as a qualified fellow eye; in this case, the Central Image Reading Center confirmed selection of the study eye. Not all subjects had a qualified fellow eye with prior treatment for PDR (Proliferative Diabetic Retinopathy).
  Participants
    Yes: number analyzed (Participants) | 13 | 20 | 22 | 55
    Yes | 1 | 2 | 5 | 8
    No: number analyzed (Participants) | 13 | 20 | 22 | 55
    No | 12 | 18 | 17 | 47
Diabetic Retinopathy Severity Scale Score in Study Eye [Mean (Standard Deviation); unit: units on a scale] — Grading will follow Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) criteria.
  DRSS grades ranging from 10-85 will be converted to an ordinal score ranging from 1-11.
  ETDRS DRSS Level 10 = No retinopathy ETDRS DRSS Level 20 = Very mild NPDR ETDRS DRSS Level 35 = Mild NPDR ETDRS DRSS Level 43 = Moderate NPDR ETDRS DRSS Level 53 = Severe NPDR ETDRS DRSS Level 61 = Mild PDR ETDRS DRSS Level 65 = Moderate PDR ETDRS DRSS Level 71-75 = High-Risk PDR ETDRS DRSS Level 81-85 = Advanced PDR
  units on a scale | 4.8 (0.70) | 4.9 (0.70) | 4.9 (0.68) | 4.9 (0.69)
Best-Corrected Visual Acuity in Study Eye, Letters [Mean (Standard Deviation); unit: letter score] | 82.4 (5.41) | 82.2 (6.40) | 83.5 (6.33) | 82.7 (6.06)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With an Improvement in Study Eye Severity of Diabetic Retinopathy (DR) (ETDRS DR Severity Score or DRSS) of ≥ 2 Steps
Description: Change from baseline to Week 48 in Diabetic Retinopathy Severity Scale Score in Study Eye by visit in the modified intent-to-treat population.
  ETDRS DR severity levels 10-85; ETDRS Steps 1-12
Time Frame: Baseline to Week 48
Population: The modified intent-to-treat population consisted of all enrolled subjects who received at least 1 dose of study medication and was the population used for the efficacy population.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Razuprotafib 15mg Twice Daily | Razuprotafib 15mg Daily | Placebo Twice Daily
Number analyzed (Participants) | 52 | 52 | 53
Number analyzed (eyes) | 52 | 52 | 53
eyes | 0 | 5 | 2
Statistical Analysis 1: Comparison: Razuprotafib 15mg Twice Daily; The primary hypotheses tested was that razuprotafib 15 mg twice daily and razuprotafib 15 mg once daily will be superior to placebo in the improvement of diabetic retinopathy as measured by the Early Treatment Diabetic Retinopathy Study severity scale change from baseline at 48 weeks; Test type: Superiority — The primary hypotheses was tested in the modified intent-to-treat population using a Fisher's Exact Test with a 2-sided 5% significance level. razuprotafib 15 mg twice daily was tested first. If this was found to be statistically significant, then razuprotafib 15 mg once daily will be tested for statistical significance, at the same significance level; p = 0.495, Fisher Exact — Missing data was imputed using last observation carried forward; baseline values were not carried forward

2. Secondary Outcome: Summary of Subjects With a Worsening in the Study Eye DRSS of ≥ 2 Steps at Week 48
Description: Worsening of Diabetic Retinopathy Severity Score (DRSS) severity of ≥ 2 steps in study eyes at Week 48 (compared to placebo group)
  Grading will follow Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) criteria.
  DRSS grades ranging from 10-85 will be converted to an ordinal score ranging from 1-11.
  ETDRS DRSS Level 10 = No retinopathy ETDRS DRSS Level 20 = Very mild NPDR ETDRS DRSS Level 35 = Mild NPDR ETDRS DRSS Level 43 = Moderate NPDR ETDRS DRSS Level 53 = Severe NPDR ETDRS DRSS Level 61 = Mild PDR ETDRS DRSS Level 65 = Moderate PDR ETDRS DRSS Level 71-75 = High-Risk PDR ETDRS DRSS Level 81-85 = Advanced PDR
Time Frame: Baseline to Week 48
Population: as for outcome 1
Measure: Count of Units; unit: study eyes
Units Other Than Participants: study eyes
Arm/Group | AKB-9778 15mg Daily | AKB-9778 15mg Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 52 | 52 | 53
Number analyzed (study eyes) | 52 | 52 | 53
study eyes | 5 | 6 | 4

3. Secondary Outcome: Mean Change From Baseline in DRSS in the Study Eye at Week 48
Description: Mean change from baseline in Diabetic Retinopathy Severity Score (DRSS) in the study eye at week 48. Note: Observed values at Week 48 instead of change from baseline values at Week 48 were analyzed
  Grading will follow Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) criteria.
  DRSS grades ranging from 10-85 will be converted to an ordinal score ranging from 1-11.
  ETDRS DRSS Level 10 = No retinopathy ETDRS DRSS Level 20 = Very mild NPDR ETDRS DRSS Level 35 = Mild NPDR ETDRS DRSS Level 43 = Moderate NPDR ETDRS DRSS Level 53 = Severe NPDR ETDRS DRSS Level 61 = Mild PDR ETDRS DRSS Level 65 = Moderate PDR ETDRS DRSS Level 71-75 = High-Risk PDR ETDRS DRSS Level 81-85 = Advanced PDR
Time Frame: Week 48
Population: Modified Intent-to-Treat Population With at Least 1 Scheduled Post-Baseline Measure (LOCF)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AKB-9778 15mg Daily | AKB-9778 15mg Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 52 | 52 | 53
score on a scale | 5.0 (1.15) | 4.9 (1.55) | 4.8 (1.35)

4. Secondary Outcome: Summary of Subjects With an Improvement or Worsening in the Study Eye DRSS of ≥ 3 Steps at Week 48.
Description: Summary of subjects with an improvement or worsening in the study eye Diabetic Retinopathy Severity Score (DRSS) of ≥ 3 steps at Week 48 (compared to placebo)
  Grading will follow Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) criteria.
  DRSS grades ranging from 10-85 will be converted to an ordinal score ranging from 1-11.
  ETDRS DRSS Level 10 = No retinopathy ETDRS DRSS Level 20 = Very mild NPDR ETDRS DRSS Level 35 = Mild NPDR ETDRS DRSS Level 43 = Moderate NPDR ETDRS DRSS Level 53 = Severe NPDR ETDRS DRSS Level 61 = Mild PDR ETDRS DRSS Level 65 = Moderate PDR ETDRS DRSS Level 71-75 = High-Risk PDR ETDRS DRSS Level 81-85 = Advanced PDR
Time Frame: Baseline to Week 48
Population: as for outcome 1
Measure: Count of Units; unit: study eyes
Units Other Than Participants: study eyes
Arm/Group | AKB-9778 15mg Daily | AKB-9778 15mg Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 52 | 52 | 53
Number analyzed (study eyes) | 52 | 52 | 53
study eyes
  Worsening ≥3 steps | 3 | 4 | 3
  Improvement ≥3 steps | 0 | 0 | 0

5. Secondary Outcome: Subjects With Criterion Step Improvement in DRSS at Week 48/EOT (>=2 Steps Improvement in the Study Eye for Patients With Non-qualified Fellow Eye and >=3 Steps Improvement on the Person Scale for Patients With Qualified Fellow Eyes)
Description: Subjects with Criterion Step Improvement in Diabetic Retinopathy Severity Score (DRSS) at Week 48/EOT (>=2 Steps Improvement in the Study Eye for Patients with Non-qualified Fellow Eye and >=3 Steps Improvement on the Person Scale for Patients with Qualified Fellow Eyes).
  Grading will follow Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) criteria.
  DRSS grades ranging from 10-85 will be converted to an ordinal score ranging from 1-11.
  ETDRS DRSS Level 10 = No retinopathy ETDRS DRSS Level 20 = Very mild NPDR ETDRS DRSS Level 35 = Mild NPDR ETDRS DRSS Level 43 = Moderate NPDR ETDRS DRSS Level 53 = Severe NPDR ETDRS DRSS Level 61 = Mild PDR ETDRS DRSS Level 65 = Moderate PDR ETDRS DRSS Level 71-75 = High-Risk PDR ETDRS DRSS Level 81-85 = Advanced PDR
Time Frame: Treatment Period - 12 months (48 weeks)
Population: Modified Intent-to-Treat Population with at least 1 scheduled Post-Baseline Measure (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | AKB-9778 15mg Daily | AKB-9778 15mg Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 52 | 52 | 53
Participants | 0 | 5 | 1

6. Secondary Outcome: Subjects With Criterion Step Improvement in DRSS at Week 48/EOT (>=2 Steps Improvement in the Study Eye for Patients With Non-qualified Fellow Eye and >=3 Steps Improvement on the Binocular Scale for Patients With Qualified Fellow Eyes)
Description: Subjects With Criterion Step Improvement in Diabetic Retinopathy Severity Score (DRSS) at Week 48/EOT (>=2 Steps Improvement in the Study Eye for Patients With Non-qualified Fellow Eye and >=3 Steps Improvement on the Binocular Scale for Patients With Qualified Fellow Eyes).
  Grading will follow Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) criteria.
  DRSS grades ranging from 10-85 will be converted to an ordinal score ranging from 1-11.
  ETDRS DRSS Level 10 = No retinopathy ETDRS DRSS Level 20 = Very mild NPDR ETDRS DRSS Level 35 = Mild NPDR ETDRS DRSS Level 43 = Moderate NPDR ETDRS DRSS Level 53 = Severe NPDR ETDRS DRSS Level 61 = Mild PDR ETDRS DRSS Level 65 = Moderate PDR ETDRS DRSS Level 71-75 = High-Risk PDR ETDRS DRSS Level 81-85 = Advanced PDR
Time Frame: Treatment Period - 12 months (48 weeks)
Population: Modified Intent-to-Treat Population with at least 1 scheduled Post-Baseline Measure (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | AKB-9778 15mg Daily | AKB-9778 15mg Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 52 | 52 | 53
Participants | 0 | 5 | 1

7. Secondary Outcome: Summary of Patients Developing Center-involved DME or PDR or PDR-related Outcomes During Treatment Period Based on Clinical Data.
Description: Summary of patients developing center-involved Diabetic Macular Edema (DME) or Proliferative Diabetic Retinopathy (PDR) or PDR-related outcomes during treatment period based on Clinical Data. Based on either clinical data or central image reading center evaluation.
Time Frame: Treatment Period - 12 months (48 weeks)
Population: mITT Population With ≥1 Scheduled Post-Baseline Measure (LOCF)
Measure: Count of Units; unit: study eyes
Units Other Than Participants: study eyes
Arm/Group | AKB-9778 15mg Daily | AKB-9778 15mg Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 52 | 52 | 53
Number analyzed (study eyes) | 52 | 52 | 53
study eyes | 12 | 10 | 10

8. Secondary Outcome: Summary of Subjects Developing Center-involved DME or PDR or Worsening of >=2 Steps DRSS at Week 48 Based on Central Image Reading Center Evaluation
Description: Summary of Subjects Developing Center-involved Diabetic Macular Edema (DME) or Proliferative Diabetic Retinopathy (PDR) or Worsening of >=2 Steps Diabetic Retinopathy Severity Scale (DRSS) at Week 48 Based on Central Image Reading Center Evaluation - Study Eyes
  Grading will follow Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) criteria.
  DRSS grades ranging from 10-85 will be converted to an ordinal score ranging from 1-11.
  ETDRS DRSS Level 10 = No retinopathy ETDRS DRSS Level 20 = Very mild NPDR ETDRS DRSS Level 35 = Mild NPDR ETDRS DRSS Level 43 = Moderate NPDR ETDRS DRSS Level 53 = Severe NPDR ETDRS DRSS Level 61 = Mild PDR ETDRS DRSS Level 65 = Moderate PDR ETDRS DRSS Level 71-75 = High-Risk PDR ETDRS DRSS Level 81-85 = Advanced PDR
Time Frame: Treatment Period - 12 months (48 weeks)
Population: Modified Intent-to-Treat Population With at Least 1 Scheduled Post-Baseline Measure (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | AKB-9778 15mg Daily | AKB-9778 15mg Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 52 | 52 | 53
Participants | 10 | 8 | 7

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Screening through the last protocol specified visit [approximately 56 weeks (Screening period up to 4 weeks, Baseline and Treatment period for 48 weeks, and Follow-up period for 4 weeks)]
Arm/Group | Razuprotafib 15mg Twice Daily | Razuprotafib 15mg Daily | Placebo Twice Daily
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55 | 1/57
Serious Adverse Events (participants affected / at risk) | 8/55 | 6/55 | 5/57
Other Adverse Events (participants affected / at risk) | 55/55 | 55/55 | 57/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Razuprotafib 15mg Twice Daily (N=55) | Razuprotafib 15mg Daily (N=55) | Placebo Twice Daily (N=57)
Osteomyelitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Burn infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diabetic gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Razuprotafib 15mg Twice Daily (N=55) | Razuprotafib 15mg Daily (N=55) | Placebo Twice Daily (N=57)
Nasopharyngitis (Infections and infestations) | 5 (5) | 4 (5) | 8 (11)
Urinary tract infection (Infections and infestations) | 7 (8) | 4 (4) | 2 (2)
Influenza (Infections and infestations) | 3 (3) | 5 (5) | 4 (4)
Sinusitis (Infections and infestations) | 2 (2) | 3 (3) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 1 (1) | 5 (5)
Bronchitis (Infections and infestations) | 4 (4) | 2 (2) | 0 (0)
Localized infection (Infections and infestations) | 0 (0) | 3 (3) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Osteomyelitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Diabetic retinal oedema (Eye disorders) | 7 (10) | 8 (10) | 7 (8)
Retinal neovascularisation (Eye disorders) | 2 (3) | 4 (6) | 7 (10)
Vitreous floaters (Eye disorders) | 2 (2) | 2 (5) | 4 (5)
Dry eye (Eye disorders) | 1 (1) | 2 (4) | 4 (8)
Eye pain (Eye disorders) | 0 (0) | 3 (4) | 3 (3)
Visual acuity reduced (Eye disorders) | 1 (3) | 3 (3) | 1 (1)
Vitreous detachment (Eye disorders) | 1 (2) | 1 (1) | 3 (4)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 3 (3) | 2 (2)
Conjunctival haemorrhage (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Ocular hyperaemia (Eye disorders) | 1 (2) | 2 (7) | 1 (1)
Visual impairment (Infections and infestations) | 2 (3) | 1 (1) | 1 (1)
Cataract nuclear (Eye disorders) | 1 (2) | 0 (0) | 2 (4)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 2 (3)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 2 (3)
Macular fibrosis (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Cataract cortical (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract subcapsular (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pruritis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Iris adhesions (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Presbyopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Pterygium (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Pupillary reflex impaired (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal cyst (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal exudate (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hyphaema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are not employed by the organization sponsoring the study

DOCUMENTS (2):
  • Study Protocol (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT03197870/Prot_001.pdf
  • Statistical Analysis Plan (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/70/NCT03197870/SAP_002.pdf